CLINICAL TRIAL: NCT03328286
Title: Improving Integration of Mentally Burdened Young Adults in the Labour Market
Acronym: inklusiv
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zurich University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Filomena Sabatella, MSc, Zurich University of Applied Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-00936
Record Dates: First submitted 2017-09-26; First posted 2017-11-01 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Mental Disorder
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Weekly group meeting w/psychotherapist (Experimental): All the participants fulfilling the eligibility criteria are asked to take part in an additional Intervention. The Intervention is a weekly group Meeting with a psychotherapist to discuss issues or Problems the Group members have
  Interventions: Behavioral: Weekly group meeting w/psychotherapist

INTERVENTIONS:
Behavioral: Weekly group meeting w/psychotherapist — Introduce a Psychotherapist in a work Integration program to further support Young adults in Job search and at the same time offering psychotherapeutic counselling. The participants will have a weekly meeting lasting 1.5 hour and additionally the can have 5 private counselling sessions with the psychotherapist if they wish

SUMMARY:
Young adults who do not successfully transition from compulsory education to upper secondary level are at increased risk of developing mental illness, as compared with their working peers. The causality is unclear: they are either unable to find a job due to a pre-existing mental illness, or their failure in finding a job has contributed to the mental illness.

The Zurich University of Applied Sciences has developed an innovative intervention that includes psychotherapeutic support in a work integration programme. Recognising and treating mental illness early increases the chances of a successful transition to the labour market.

DETAILED DESCRIPTION:
Unemployed young people with severe psychological impairments often find no training or workplace, despite the support of various existing services. Many of these young people suffer from a mental illness, but they are often neither diagnosed nor treated. In Switzerland, this is reflected in the increasing number of young people who receive a disability pension. To make matters worse, young people often do not use the necessary psychotherapeutic treatment. An explanation for this may be the fear of being stigmatized or the lack of insight that help is needed al all. A group of researchers has analyzed the dossiers of 400 young people who were given a disability pension 2010 and 2013 due to mental problems. They have found that the consultation often took place before the 23rd year of age and in 84% of the cases whole disability pensions were given. In the analysed cases only 14% had completed vocational training. The authors propose various measures, including prioritizing the completion of a professional apprenticeship, a systematic interdisciplinary assessment, a joint, longer-lasting integration management, as well as early detection and intervention in psychological disorders in school and vocational training. Our intervention meets these requirements. Together with lifetime health, a provider work working integrations programs, we have developed a low-threshold psychotherapeutic offer in addition to the existing work integration program. With this intervention we hope to reach the following goals. First: Facilitate the transition into a professional apprenticeship by increasing work ability and other variables. Secondly, the integration and cooperation of a psychotherapist in the work integration program allows for a systematic interdisciplinary assessment; third, the support of a psychotherapist offers a joint, longer-lasting integration management.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 to 25
* Participation in work integration programme "Lifetimehealth"

Exclusion Criteria:

* Insufficient knowledge of German
* Participant is under guardianship which doesn't allow legal capacity to act

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Work Ability | Up to 2 years
  Increase in work ability of participants, measured with the Work Ability Index. The Work Ability Index (WAI) is an instrument used in occupational health care and research to assess work ability of workers during health examinations and workplace surveys. The purpose of WAI is to help define necessary actions to maintain and promote work ability. The scoring system of the questionnaire categorises work ability, with recommendations for action provided for each category. Appropriate action can then be taken to prevent declining work ability.Each answer has a different score, with users calculating their total points to determine their final score. The minimum is 7, the maximum is 49. The four categories of scores and the objectives of the measures to be taken are as follows:
  * 7-27 points (bad) - restore work ability;
  * 28-36 points (moderate) - improve work ability;
  * 37-43 points (good) - support work ability;
  * 44-49 points (very good) - support work ability.

SECONDARY OUTCOMES:
Change in Self-esteem | Up to 2 years
  Increase in self-esteem of participants, measured with the Rosenberg Self-esteem Scale (SES). The SES is a 10-item scale that measures global self-worth by measuring both positive and negative feelings about the self.
  Scores are calculated as follows:
  •For items 1, 2, 4, 6, and 7: Strongly agree = 3 Agree = 2 Disagree = 1 Strongly disagree = 0
  •For items 3, 5, 8, 9, and 10 (which are reversed in valence): Strongly agree = 0 Agree = 1 Disagree = 2 Strongly disagree = 3
  The scale ranges from 0-30. Scores between 15 and 25 are within normal range; scores below 15 suggest low self-esteem.

CONTACTS AND LOCATIONS:
Overall Officials: Agnes von Wyl, Prof, Principal Investigator — University of applied sciences
Locations (1):
- Toni Areal, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sabatella F, von Wyl A. Improving Work Ability of Mentally Burdened Emerging Adults in Vocational Integration Programs: A Study Protocol. Front Psychol. 2019 Jun 19;10:1391. doi: 10.3389/fpsyg.2019.01391. eCollection 2019. PMID 31275206